CLINICAL TRIAL: NCT03785639
Title: Factors Contributing to Single and Dual Task Performance of Four Square Step Tests in the Healthy Middle Age Group
Brief Title: Factors Contributing to Single and Dual Task Performance of Four Square Step Tests
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Suat EREL, Principal Investigator, Pamukkale University
Other Study IDs: 60116787-020/71491
Record Dates: First submitted 2018-12-18; First posted 2018-12-24 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Aging
Keywords: balance; dual task; Four Square Step Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are many tests that evaluate fall and balance. As a clinical test, the Four Square Step Test (FSST)Test is reliable, valid, easy to score, quick to administer, requires little space, and needs no special equipment. It is unique in that it involves stepping over low objects (2.5cm) and movement in 4 directions. FSST was developed in 2002 to measure the rapid stepping that is often required when changing direction and avoiding obstacles while walking. The FSST requires a stopwatch and four single point sticks. Using the sticks resting flat on the floor to form a cross, the subject starts in one square and steps in one direction into each of the four squares and then reverses direction back to the start. The FSST is unique in that it challenges motor planning, sequencing and recall, whilst simultaneously providing clinicians with the opportunity to measure and observe a person's clearance of low obstacles at speed. The ability to clear the trail leg when stepping over an obstacle has been shown to be reduced in healthy populations. Dual task is simultaneous performance of two tasks that can be performed independently, measured separately and with different goals. Individuals have difficulties in performing two tasks together. When two tasks are performed at the same time, deterioration in performance of one or both is called dual task interference. This occurs when task requirements exceed the capacity. Age, walking speed, lower extremity muscle strength and cognitive status are factors that contribute to the dual task. In addition, prioritizing the motor or cognitive task in a dual task affects the dual task performance. Knowing these factors and improving some of them can help to create training programs designed to improve the dual task performance of individuals. There are several studies investigating factors contributing to dual task performance that focus on balance in the elderly. However, the studies including middle age group are limited. There are no studies evaluating the factors contributing to the single and dual task performance of FSST in the literature. In this study, it is aimed to explain the factors related to motor and cognitive functions to the single and dual task performance of FSST.

DETAILED DESCRIPTION:
Participants: Healthy middle age group (50-65 years) Method: Demographic information of all participants (age, gender, body mass index), educational level (primary, undergraduate, graduate), history of falling (at least in 6 months), comorbidities (hypertension, diabetes, kidney diseases, etc.), drug using (how many per day, which one) to be examined by questionnaire and also visual impairment, the use of glasses will be recorded. Motor skills of participants; muscle strength, range of motion (ROM), gait speed (14m), Functional Reach Test will be evaluated. The Mini Mental Test and the Stroop test will be used to evaluate cognitive skills. Single and dual task performance will be evaluated by FSST.

The participants performed the FSST;

1. FSST single: This test is consist of only FSST.
2. FSST motor: FSST is combined with a motor task (carrying a cup of water)
3. FSST cognitive: FSST is combined with a cognitive task (auditory N-back test) As prioritization affects dual task performance, in this study the prioritization will be used in dual task's evaluation. Therefore the dual task will be perform as;

1-With no prioritization 2-With prioritization (focus on balance task) 3-With prioritization (focus on cognitive task) 4-With prioritization (focus on motor task) Note: Balance task is FSST. Cognitive task is auditory N-back test. Motor task is carrying a cup of water.

Statistical Analyses:

The data will be analyzed with Statistical Package for the Social Sciences (SPSS) 21.0 package program. Descriptive statistical information will be given as mean (X) ± standard deviation (X ± SD) and minimum (min), maximum (max) frequency (f) and percentage (%). The variables will be tested for normality using the Kolmogorov-Smirnov test. When the parametrical test assumptions are obtained, the correlation between the FSST single, FSST motor and FSST cognitive is evaluated by Pearson Correlation Analysis, if the parametrical test assumptions are not obtained, Spearman Correlation Analysis will be used. Multiple linear regression analysis will be applied to determine which potential factor is effective in performance in each FSST test. As a result of the power analysis using the effect size value in the reference study for the study, it was calculated that 85% power could be obtained at 95% confidence level when at least 60 people.

ELIGIBILITY:
Inclusion Criteria:

* At least to graduate from primary school or ability to read and write
* Mini mental test score> 24
* Functional reach test score≥15 cm
* Ability to walking independently in the community

Exclusion Criteria:

* Living in nursing home
* Presence of central nervous system disease (dementia, Parkinson's disease, stroke, etc.)
* Polypharmacy (more than 6 medications per day)
* Presence of hearing impairment that cannot be resolved by hearing devices and presence visual impairment that cannot be resolved by hearing aids.
* Presence of musculoskeletal injuries or impairments (NEH limitation, muscle weakness, etc.), which may affect the performance in physical tests

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty healthy active (joining social activities, sports and artistic activities etc.) participants (men and women) between the ages of 50-65 will be included in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | 20 minutes
  Grip strength and muscle strength of low extremities will be evaluated with using hand-held dynamometer. The measured value will be recorded in newton.
Range of motion | 10 minutes
  Range of motions of hip, knee and ankle will be assessed by goniometer.
Gait speed | 2 minutes
  Gait speed will be evaluated on a flat surface and at a distance of 14 meters. The walking speed will be recorded in m/sec.
Functional ReachTest | 2 minutes
  The FRT assesses limits of stability by measuring the maximum distance that an individual can reach forward while standing in a fixed position. A 122 cm ruler will be fastened to the wall with tape at the height of the subject's acromion process. The subject will be instructed to make a fist and raise the arm to 90 degrees of shoulder flexion. An initial measurement will be record at the position of the subject's third metacarpal. The subject will be instructed to reach as far forward as possible while keeping the fist parallel and level with the ruler and without taking a step or touching the wall.
Stroop Test | 10 minutes
  This test evaluate cognitive abilities. the Stroop Test is a useful measuring tool for especially the fields of psychiatry, neurology, neurosurgery, and clinical psychology and for the basic science field of experimental psychology. The test is used to evaluate cognitive processes such as frontal lobe functions and attention, information processing periods.
Four Square Step Test (FSST) | 20 minutes
  FSST is designed for assessing balance. The participants will be asked to stand in square number 1 facing square number 2 and to step clockwise forward, then right, backward and left, then anticlockwise right, forward and left and finally backward. The stopwatch will start when the first foot contacted the floor in square 2 and will finish when the last foot came back to touch the floor in square 1. Single and dual task performance will be evaluated by FSST.
  The participants performed the FSST; FSST single: This test is consist of only FSST. FSST motor: FSST is combined with a motor task (carrying a cup of water) FSST cognitive: FSST is combined with a cognitive task (auditory N-back test) As prioritization affects dual task performance, in this study the prioritization will be used in dual task's evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Emel TAŞVURAN HORATA, MSc, Principal Investigator — Principal Investigator
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yogev-Seligmann G, Rotem-Galili Y, Mirelman A, Dickstein R, Giladi N, Hausdorff JM. How does explicit prioritization alter walking during dual-task performance? Effects of age and sex on gait speed and variability. Phys Ther. 2010 Feb;90(2):177-86. doi: 10.2522/ptj.20090043. Epub 2009 Dec 18. PMID 20023000